CLINICAL TRIAL: NCT04453865
Title: Empowering Anxious Parents to Manage Child Avoidance Behaviors: A Randomized Trial of a Single-Session Intervention Targeting Parent Accommodation
Brief Title: Empowering Anxious Parents to Manage Child Avoidance Behaviors
Acronym: EMPOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor of Psychology, Stony Brook University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB2020-00069
Record Dates: First submitted 2020-05-28; First posted 2020-07-01 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Parenting; Accommodation; Online Intervention; Single Session Intervention
MeSH Terms: conditions — Anxiety Disorders | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized via Qualtrics (1:1 allocation ratio) to either the Online Resources and Referrals (ORR) and the Parent Accommodation SSI or ORR alone and delayed SSI access. Those in the experimental condition (ORR+immediate SSI) will also complete immediate post-SSI questionnaires. Two weeks later, all parents-regardless of condition-will complete the 2-week follow up questionnaires. Parents in the ORR+delayed SSI condition will then be invited to complete the accommodation SSI and immediate post-SSI questionnaires. Thus, all participants will receive the accommodation SSI and complete immediate post-SSI questionnaires, either immediately or at 2-week follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project EMPOWER (Experimental): Project EMPOWER is a web-based, self-administered SSI for parents that takes about 30 minutes to complete. The program includes 5 elements, based on current best-practices in SSI design (Schleider, Dobias, Sung, & Mullarkey, 2020) and existing interventions targeting accommodation (Lebowitz & Omer, 2014): (1) an introduction to the program's rationale; (2) psychoeducation around child anxiety and avoidance, along with how parental accommodation can inadvertently maintain child anxiety; (3) information on how parents can better identify children's patterns of avoidance and encourage brave behavior instead; (4) facilitating parents' creation of an "action plan" for promoting brave behavior and reduce avoidance in their own child; (5) a vignette exercise in which parents read about another family's difficulty managing their child's anxiety; parents identify the elements of the anxiety cycle and provide possible solutions to these parents based on what they learned.
  Interventions: Behavioral: Project EMPOWER
- Online Resources and Referrals (ORR) (Other): Online Resources and Referrals (ORR) is an information sheet containing materials about the nature of child anxiety and a list of national resources related anxiety treatment. ORR does not include any psychoeducational components regarding parental accommodation.
  Interventions: Other: Online Resources and Referrals

INTERVENTIONS:
Behavioral: Project EMPOWER — Project EMPOWER is a web-based, self-administered SSI for parents that takes about 30 minutes to complete
  Arms: Project EMPOWER
Other: Online Resources and Referrals — Information sheet containing materials about the nature of child anxiety and a list of national resources related anxiety treatment.
  Other Names: ORR
  Arms: Online Resources and Referrals (ORR)

SUMMARY:
Efforts to develop and disseminate evidence based practices (EBPs) for youth anxiety have made great strides. Still, up to 82.2% of youth who need mental health treatment for anxiety never access care or drop out prematurely; commonly cited barriers to treatment are shortage of care, transportation limitations, financial burden, and gatekeeping behaviors by caretakers. As such, there is great need for accessible, scalable interventions that can ameliorate the global burden of youth anxiety, including those that help prevent the onset of anxiety in high-risk children. Single session interventions (SSIs), which have prevented and reduced child anxiety across numerous trials to date, may offer a promising solution, given their potential disseminability and cost-effectiveness. The proposed randomized trial will evaluate the effects of a novel, web-based, self-guided SSI designed to systematically reduce parent accommodation: a parenting behavior identified as a strong risk factor for anxiety in offspring. Study aims will be three-fold: (1) to examine the SSI's direct effects on parental accommodation, relative to an information-only control; (2) to assess the SSI's immediate effects on parents' perceived ability to help their children manage distressing situations; and (3) to evaluate the SSI's feasibility and acceptability. We will recruit parents reporting elevated anxiety levels, as children of anxious parents are at particular risk for developing anxiety symptoms themselves. Results may suggest a promising approach to preventing anxiety in at-risk children.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common, debilitating forms of childhood psychopathology, affecting 8.3-27.0% of youth before the age of 18. Child anxiety increases risk for psychiatric comorbidities across the lifespan) creates significant burdens for caregivers, and carries societal costs. Although numerous interventions have been developed to treat youth anxiety disorders, up to 82.2% of US youth with anxiety will not receive adequate care. Several reasons may explain this discrepancy, including the length and cost of existing evidence-based interventions (EBIs) and limited accessibility for families in need.

Single-session interventions (SSIs) may offer one potential solution to this gap in care. SSIs include core components of comprehensive EBIs delivered succinctly to improve the odds of access and completion. In a recent meta-analysis of 50 RCTs, SSIs reduced youth mental health problems of multiple disorders, with SSIs targeting child anxiety producing the largest effects (mean g = 0.58). Thus, well-targeted SSIs may offer cost-effective additions or alternatives to traditional care for anxiety in youth. However, most existing SSIs for child anxiety target populations already experiencing clinical distress, and a need remains for options that may prevent anxiety in vulnerable children. Given that family factors play a crucial role in the etiology of child anxiety, SSIs targeting parents and their interactions with offspring offer a novel approach to preventing youth anxiety. Thus, the aim of this project is to test the acceptability and short-term effects of a novel, web-based SSI targeting parental accommodation: a well-established, potentially modifiable risk factor for child anxiety. Results may reveal a promising, targeted approach to scalable child anxiety prevention.

Parental Accommodation as a Modifiable Intervention Target. Parent accommodation refers to changes in caregiver behaviors that facilitate or maintain their child's avoidance or anxiety. Examples include modifying family routines (i.e., staying home from work to alleviate a child's fear of separating) or directly participating in a child's avoidance strategies (i.e., keeping a child home from school). Parent accommodation reduces immediate distress but maintains long-term avoidance of feared stimuli or situations and high levels of parent accommodation are associated with anxiety problems in offspring. Parent accommodation is further maintained by caregiver factors, including parental anxiety and tolerance for distress. For instance, accommodation is greater among parents reporting higher distress about their child's anxiety symptoms and perceptions that anxiety exposure is harmful for youth.

Research shows that parent accommodation can be systematically reduced via psychosocial intervention, and interventions targeting accommodation have helped mitigate child anxiety. Translating core components of existing interventions that target parental accommodation into briefer, self-administered SSIs (i.e., those that do not involve a trained therapist) may improve families' access to empirically-driven supports for child anxiety. It may also enhance the implementation of mental health interventions by lay providers who frequently interact with children (e.g. teachers and pediatricians). Thus, the goal of this project is to test a web-based, self-guided SSI targeting parental accommodation. Parent participants will be randomized to either (a) Online Resources and Referrals (ORR) + parent accommodation SSI, or (b) ORR alone and delayed SSI access. We predict that parents will report larger declines in accommodation in the ORR+Accommodation SSI group, relative to the ORR + delayed SSI access group, from baseline to 2-week follow-up. We also predict that parents will perceive significant pre-to immediate-post-SSI increases in their ability to help their child manage distressing situations. Finally, we predict that participants will find the SSI to be acceptable.

ELIGIBILITY:
Inclusion Criteria:

1. Report subclinical or greater anxiety symptoms, per a score of 40 or higher on the Penn State Worry Questionnaire (PSWQ)
2. Have at least one child between the ages of 4-10 years old
3. Live in the United States (US)

Exclusion Criteria:

1. Participant is non-English speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Family Accommodation Scale | Change from Baseline Accommodation at 2-week follow up
  Family Accommodation Scale is a 9-item measure designed to assess the extent a caregiver accommodate a child's anxiety symptoms; example questions include: "how often did you assist your child in avoiding things that might make him/her more anxious?" and "have you modified your family routine because of your child's symptoms?" Items are rated from 0 (never) to 4 (daily). Scores range from 0-36 with higher scores indicating more frequent parental accommodation.
Perceived pre-to-post SSI change | Immediately after the SSI
  This single-item measure assesses participants' perceived change in their ability to help their children manage distressing situations from pre- to post-SSI: "compared to before you completed this program, how prepared do you feel to help your child manage distressing situations?" Parents in both groups will rate this question on a 5-point scale of 1 (much less able to help child manage distressing situations) to 5 (much more able to to help child manage distressing situations).

SECONDARY OUTCOMES:
Program Feedback Scale | Immediately after the SSI
  The program feedback scale asks participants to rate 7 statements regarding acceptability and feasibility; note whether they would recommend this activity to others; and share what they liked and would change about the SSI. The 7 statements are rated from 0 (Really Disagree) to 5 (Really Agree). Total score ranges from 0 to 35, with higher scores indicating a more positive program evaluation.
Penn State Worry Questionnaire | Baseline
  16 item self-report questionnaire that asks individuals to rate how typical worry-related problems are for them, from 1 (not at all typical) to 5 (very typical). Scores range from 16-80; higher scores indicate more severe worry.
Coping with Children's Negative Emotions Scale | Baseline
  Coping with Children's Negative Emotions Scale measures parents' reactive emotions to their child's negative affect in distressing situations. Six subscales exist, but only the "distress reactions" domain, reflecting parental distress in the context of child negative affect, will be used. Participants rate 12 questions from 1 (very unlikely) to 7 (very likely). Score ranges from 12-84; higher numbers indicate more distress.
Revised Children's Anxiety and Depression Scale | Baseline
  25 item measure assessing child's symptoms of anxiety and depression. Each question is rated on a 4-point scale from 0 (Never) to 3 (Always). Total score ranges from 0 to 75 with higher scores indicating higher levels of psychopathology
Barriers to Access to Care Evaluation | Baseline
  30 item self-report questionnaire that asks about barriers they faced in getting professional care for a mental health problem on a scale of 0 (not at all) to 3 (a lot). Scores range from 0 to 90; higher scores indicate a higher number of barriers.
Adult Measure of Behavioral Inhibition | Baseline
  16 item measure assessing one's temperamental tendency to respond to social novelty and risk stimuli, with inhibition and avoidance. Each question is rated on a 3 point scale from 0 (no/hardly ever) and 2 (yes/most of the time). Total score ranges from 0 to 32 with a higher scores indicating a greater degree of inhibition.
Short Behavioral Inhibition Questionnaire | Baseline
  14-item parent rated scale measuring temperamental characteristics referring to shyness, fearfulness, and withdrawal in young, preschool children. Each question is rated on a 7-point scale from 1 (Hardly Ever) to 7 (Almost Always). Total score ranges from 14 to 98, with higher scores indicating a greater degree of inhibition
Ruminative Response Scale | Baseline
  22 item questionnaire measuring two aspects of rumination: brooding and reflective pondering. Each question is rated on a 4-point scale from 1 (almost never) and 4 (almost always). Total score ranges from 22 to 88 with a higher score indicating higher ruminative tendencies.
Distress Tolerance Scale | Change from Baseline Coping at 2-week follow up
  16 item measure assessing the extent to which one experiences and withstand distressing emotional states. Each item is rated on a 5-point Likert scale from 1 (strongly agree) and 5 (strongly disagree). Total score ranges from 16 to 80 with a higher score indicating higher levels of distress tolerance.
Co-Rumination Questionnaire | Baseline
  27-item self-report inventory that measures the extent to which one co-ruminates with others. For brevity, the survey has been modified to consist of 8 items that range from 1 (Not at all true) to 5 (really true). Total score ranges from 8 to 40 with a higher score indicating higher levels of co-rumination.
Patient Reported Outcomes Measurement Information System-Depression Short | Baseline
  8 item self-report measure of depression. The questions are rated on a 5-point scale ranging from 1 (never) to 5 (always). Scores range from 8 to 40m higher scores indicating higher levels of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beecham J. Annual research review: Child and adolescent mental health interventions: a review of progress in economic studies across different disorders. J Child Psychol Psychiatry. 2014 Jun;55(6):714-32. doi: 10.1111/jcpp.12216. Epub 2014 Feb 28. PMID 24580503
- [Background] Bodden DH, Dirksen CD, Bogels SM. Societal burden of clinically anxious youth referred for treatment: a cost-of-illness study. J Abnorm Child Psychol. 2008 May;36(4):487-97. doi: 10.1007/s10802-007-9194-4. Epub 2008 Jan 23. PMID 18214667
- [Background] Copeland WE, Angold A, Shanahan L, Costello EJ. Longitudinal patterns of anxiety from childhood to adulthood: the Great Smoky Mountains Study. J Am Acad Child Adolesc Psychiatry. 2014 Jan;53(1):21-33. doi: 10.1016/j.jaac.2013.09.017. Epub 2013 Oct 12. PMID 24342383
- [Background] Costello EJ, Egger HL, Angold A. The developmental epidemiology of anxiety disorders: phenomenology, prevalence, and comorbidity. Child Adolesc Psychiatr Clin N Am. 2005 Oct;14(4):631-48, vii. doi: 10.1016/j.chc.2005.06.003. PMID 16171696
- [Background] Degnan KA, Almas AN, Fox NA. Temperament and the environment in the etiology of childhood anxiety. J Child Psychol Psychiatry. 2010 Apr;51(4):497-517. doi: 10.1111/j.1469-7610.2010.02228.x. Epub 2010 Feb 11. PMID 20158575
- [Background] Edlund MJ, Unutzer J, Curran GM. Perceived need for alcohol, drug, and mental health treatment. Soc Psychiatry Psychiatr Epidemiol. 2006 Jun;41(6):480-7. doi: 10.1007/s00127-006-0047-1. Epub 2006 Mar 25. PMID 16565918
- [Background] Kendall, P. C., Aschenbrand, S. G., & Hudson, J. L. (2003). Child-focused treatment of anxiety. Evidence-Based Psychotherapies for Children and Adolescents, 81-100.
- [Background] Lebowitz, E. R., Omer, H., Hermes, H., & Scahill, L. (2014). Parent Training for Childhood Anxiety Disorders: The SPACE Program. Cognitive and Behavioral Practice, 21(4), 456- 469. https://doi.org/10.1016/j.cbpra.2013.10.004
- [Background] Lebowitz ER, Panza KE, Su J, Bloch MH. Family accommodation in obsessive-compulsive disorder. Expert Rev Neurother. 2012 Feb;12(2):229-38. doi: 10.1586/ern.11.200. PMID 22288678
- [Background] Lebowitz ER, Scharfstein L, Jones J. Child-Report of Family Accommodation in Pediatric Anxiety Disorders: Comparison and Integration with Mother-Report. Child Psychiatry Hum Dev. 2015 Aug;46(4):501-11. doi: 10.1007/s10578-014-0491-1. PMID 25209390
- [Background] Merikangas KR, He JP, Burstein M, Swendsen J, Avenevoli S, Case B, Georgiades K, Heaton L, Swanson S, Olfson M. Service utilization for lifetime mental disorders in U.S. adolescents: results of the National Comorbidity Survey-Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2011 Jan;50(1):32-45. doi: 10.1016/j.jaac.2010.10.006. Epub 2010 Dec 3. PMID 21156268
- [Background] Mojtabai R, Olfson M, Sampson NA, Jin R, Druss B, Wang PS, Wells KB, Pincus HA, Kessler RC. Barriers to mental health treatment: results from the National Comorbidity Survey Replication. Psychol Med. 2011 Aug;41(8):1751-61. doi: 10.1017/S0033291710002291. Epub 2010 Dec 7. PMID 21134315
- [Background] Ramos-Cerqueira AT, Torres AR, Torresan RC, Negreiros AP, Vitorino CN. Emotional burden in caregivers of patients with obsessive-compulsive disorder. Depress Anxiety. 2008;25(12):1020-7. doi: 10.1002/da.20431. PMID 18833578
- [Background] Salloum A, Johnco C, Lewin AB, McBride NM, Storch EA. Barriers to access and participation in community mental health treatment for anxious children. J Affect Disord. 2016 May 15;196:54-61. doi: 10.1016/j.jad.2016.02.026. Epub 2016 Feb 10. PMID 26901657
- [Background] Schleider JL, Dobias ML, Sung JY, Mullarkey MC. Future Directions in Single-Session Youth Mental Health Interventions. J Clin Child Adolesc Psychol. 2020 Mar-Apr;49(2):264-278. doi: 10.1080/15374416.2019.1683852. Epub 2019 Dec 4. PMID 31799863
- [Background] Schleider JL, Mullarkey MC, Weisz JR. Virtual Reality and Web-Based Growth Mindset Interventions for Adolescent Depression: Protocol for a Three-Arm Randomized Trial. JMIR Res Protoc. 2019 Jul 9;8(7):e13368. doi: 10.2196/13368. PMID 31290406
- [Background] Schleider, J. L., & Weisz, J. R. (2017a). Can less be more? The promise (and perils) of single session youth mental health interventions. The Behavior Therapist, 40(7), 256-261.
- [Background] Schleider JL, Weisz JR. Little Treatments, Promising Effects? Meta-Analysis of Single-Session Interventions for Youth Psychiatric Problems. J Am Acad Child Adolesc Psychiatry. 2017 Feb;56(2):107-115. doi: 10.1016/j.jaac.2016.11.007. Epub 2016 Nov 25. PMID 28117056
- [Background] Settipani CA, Kendall PC. The Effect of Child Distress on Accommodation of Anxiety: Relations With Maternal Beliefs, Empathy, and Anxiety. J Clin Child Adolesc Psychol. 2017 Nov-Dec;46(6):810-823. doi: 10.1080/15374416.2015.1094741. Epub 2015 Dec 16. PMID 26672808
- [Background] Storch, E. A., Lehmkuhl, H., Pence, S. L., Geffken, G. R., Ricketts, E., Storch, J. F., & Murphy, T. K. (2009). Parental experiences of having a child with obsessive-compulsive disorder: Associations with clinical characteristics and caregiver adjustment. Journal of Child and Family Studies, 18(3), 249-258.
- [Background] Thompson-Hollands J, Kerns CE, Pincus DB, Comer JS. Parental accommodation of child anxiety and related symptoms: range, impact, and correlates. J Anxiety Disord. 2014 Dec;28(8):765-73. doi: 10.1016/j.janxdis.2014.09.007. Epub 2014 Sep 16. PMID 25261837
- [Derived] Sung JY, Mumper E, Schleider JL. Empowering Anxious Parents to Manage Child Avoidance Behaviors: Randomized Control Trial of a Single-Session Intervention for Parental Accommodation. JMIR Ment Health. 2021 Jul 6;8(7):e29538. doi: 10.2196/29538. PMID 34255718

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT04453865/SAP_001.pdf